CLINICAL TRIAL: NCT05740111
Title: The PREPAIRD Study: Personalized suRveillance for Early Detection and Prevention of Pancreatic cAncer in High Risk inDividuals
Brief Title: The PREPAIRD Study: Personalized Surveillance for Early Detection of Pancreatic Cancer in High Risk Individuals
Acronym: PREPAIRD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government); University of Oslo (Other); Haukeland University Hospital (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); University of Bergen (Other); Immunovia, Inc. (Industry); University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Eli Marie Grindedal, Head of Section for Hereditary Cancer, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 387940
Record Dates: First submitted 2022-10-12; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Hereditary Pancreatic Cancer
Keywords: Surveillance; Early detection; Prevention
MeSH Terms: conditions — Pancreatic carcinoma, familial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Annual surveillance — Annual surveillance includes annual MRI and/or an assessment new onset diabetes and unintended weight loss.

SUMMARY:
The objective of this national and multidisciplinary project is to establish and evaluate a personalized surveillance program (SP) for early diagnosis of pancreatic cancer (PC) and its precursors in individuals with a hereditary predisposition to the disease (High RIsk Individuals (HRI)). Patients who either carry a germline mutation in a PC susceptibility gene (CDKN2A, STK11, TP53, PRSS1), or have a strong family history of PC, will be enrolled through their genetics clinic at the university hospitals in Oslo, Bergen, Trondheim and Tromsø. Surveillance consists of annual MRI, assessment of blood glucose and lipid levels, new onset diabetes (NOD) and unintentional weight loss. Blood samples will be drawn for ctDNA-analysis (circulating tumor DNA) and the IMMrayTM PanCan-d test (a novel microarray-based diagnostic test for PC) at baseline and in those who develop lesions. The psychological burden and cost-benefit of the SP will be analyzed. The study addresses an unmet need for the care of HRI in Norway, and is expected to improve PC prognosis. It will be the first to provide evidence on the combined value of a panel of blood-borne biomarkers in surveillance, and provide morphological and molecular data on PC and (non)-neoplastic pancreatic changes in HRI.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women with a germline mutation in CDKN2A, TP53, PRSS1 or STK11
2. Men or women who are first degree relatives to a patient with pancreatic cancer (PC) in a family with Familial Pancreatic Cancer (FPC).

Exclusion Criteria: Patients undergoing active cancer treatment.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2042-12-31 (Estimated); Study Completion 2042-12-31 (Estimated)

PRIMARY OUTCOMES:
Prognosis of pancreatic cancer in patients diagnosed through the surveillance programme compared to prognosis in unscreened individuals as reported to the Cancer Registry of Norway. | Up to 20 years
  We will investigate whether 3 year, 5 year and long term survival in HRIs undergoing surveillance is improved compared to rates of survival of pancreatic cancer in the general unscreened population. Survival data for the general population will be collected from the Cancer Registry of Norway. Data on prognosis of pancreatic cancer in patients undergoing surveillance will be collected from electronic patient records, The Cancer Registry of Norway and the National Population Register.
Number of resectable cancers detected in patients diagnosed through the surveillance programme compared to the unscreened individuals as reported to the Cancer Registry of Norway. | 20 years
  We will investigate whether the number of surgically resectable cancers is higher in HRIs undergoing screening through the surveillance programme compared to pancreatic cancer diagnosed in the general population of Norway. Data on number of resectable cancers in the general Norwegian population will be collected from the Cancer Registry of Norway. Data on cancers diagnosed in the HRI will be collected from electronic patient records and The Cancer Registry of Norway.

SECONDARY OUTCOMES:
Healthcare utilization | 20 years
  Use of medication and specialist health care services. Data collected from administrative registries.
Quality of life of participants undergoing surveillance as assessed with the Hospital Anxiety and Depression Scale (HADS) | 10 years
  The quality of life of participants undergoing surveillance will be assessed with the Hospital Anxiety and Depression Scale (HADS) at baseline, after first, second and third MRI and then every three years.
Costs | Up to 20 years
  Health care utlization will be combined with Norwegian unit costs and summarized up to 20 years.
Cost-effectiveness analysis | Up to 20 years
  Differences in costs between study population and unscreened pancreatic cancer patients in the general population. Differences in survival in the PREPAIRD-study population and pancreatic cancer patients in the general population, identified from the Cancer Registry of Norway. The health outcome is identified in primary objective one. Based on difference in costs and life years, the incremental cost-effectiveness ratio will be estimated.
Quality of life of participants undergoing surveillance as assessed with the Impact of Event Scale (IES) | 10 years
  he quality of life of participants undergoing surveillance will be assessed with the Hospital Anxiety and Depression Scale (HADS) at baseline, after first, second and third MRI and then every three years.
The cancer worry of participants undergoing surveillance as assessed with the Cancer Worry Scale | 10 years
  The cancer worry of undergoing surveillance will be assessed with the Cancer Worry Scale at baseline, after first, second and third MRI and then every three years.
The general health of participants undergoing surveillance as assessed with the General Health Questionnaire | 10 years
  The cancer worry of undergoing surveillance will be assessed with the General Health Questionnaire at baseline, after first, second and third MRI and then every three years.
The psychological consequences of undergoing screening for pancreatic cancer as assessed by the Psychological Consequences of Screening questionnaire | 10 years
  The psychological consequences of undergoing screening for pancreatic cancer will be assessed with the Psychological Consequences of Screening questionnaire at baseline, after first, second and third MRI and then every three years.
The general health of participants undergoing surveillance as assessed by the Genereal Health questionnaire | 10 years
  The general health of individuals undergoing screening for pancreatic cancer will be assessed with the General Health Questionnaire at baseline, after first, second and third MRI and then every three years.
The psychological well-being of participants undergoing surveillance as assessed by the Psychological Well-being Questionnaire | 10 years
  The psychological well-being of individuals undergoing screening for pancreatic cancer will be assessed with the Psychological Well-being Questionnaire at baseline, after first, second and third MRI and then every three years.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway